CLINICAL TRIAL: NCT05443659
Title: Real-World Analysis of Remote Electrical Neuromodulation (REN) for the Acute Treatment of Migraine in Adolescence
Brief Title: Real-world Data Analysis of REN Treatment in Adolescence With Migraine
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE003
Record Dates: First submitted 2022-06-25; First posted 2022-07-05 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Migraine in Adolescence
Keywords: migraine, Headache Nerivio, REN
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Nerivio — Remote electrical neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation(CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application.

SUMMARY:
This is a Post-marketing study investigating the safety and efficacy of the REN device (Nerivio by Theranica, Israel) in adolescents with migraine. Data analysis concerning the REN treatment efficacy in terms of pain and functional disability as a standalone treatment or in combination with other medications will be performed.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, Israel) is a neuromodulation device approved by the FDA for acute treatment of migraine in patients of 12 years old and above (1-4). It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs, modulated frequency of 100-120 Hz, and up to 40 mA output current which the patient can adjust. The REN device is operated by a designated app that is downloaded to the user's phone prior first use of the Nerivio device

As part of the sign-up process to the Nerivio app, all patients accept the terms of use which specify that providing personal information is done of their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback. The app includes a secured, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability (No limitation, Some limitation, Moderate limitation, Severe limitation), and an indication of which medications, if any, were taken within that 2-hour time window.

Post-marketing surveillance is designed to assess the efficacy and safety in larger and more diverse populations and in various real-world environments and situations. As a digital therapeutic device (i.e., electroceutical), the REN device enables prospective collection of electronic patient-reported outcomes in real-world clinical practice.

Recently, Real World Evidence (RWE) papers of Nerivio usage in adults were published (5-6). these papers demonstrated the safety and efficacy of the Nerivio device in a large-scale population using the accumulated data gathered by diary within the Nerivio app.

This post-marketing RWE study investigates the efficacy of the Nerivio treatment using the following outcomes:

1. - Reduction in headache pain 2h post-treatment
2. - Improve in functional disability
3. - A standalone treatment vs combination with other therapies
4. - Safety profile (in terms of device-related adverse events)

Together, these four objectives provide a comprehensive evaluation of efficacy, drug-device interactions, dose stability, and safety, in a large real-world dataset of over XXXXX treatments in the migraine adolescent population.

ELIGIBILITY:
Inclusion Criteria:

1. - Age between 12-18 years
2. - REN user across the United States who created Nerivio account on January 1st, 2021 or later.
3. - Had at least two evaluable treatments with the Nerivio device

Exclusion Criteria:

(1) - Treatments shorter than 20 minutes

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescence (age 12-18) who suffers from migraine who are using the Nerivio device for acute treatment of migraine
Sampling Method: Probability Sample
Enrollment: 1629 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, PhD, Principal Investigator — Theranica Bio-Electronics ltd
Locations (2):
- Theranica USA Inc, Bridgewater, New Jersey, United States
- Theranica Bio-Electronics Ltd, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yarnitsky D, Dodick DW, Grosberg BM, Burstein R, Ironi A, Harris D, Lin T, Silberstein SD. Remote Electrical Neuromodulation (REN) Relieves Acute Migraine: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial. Headache. 2019 Sep;59(8):1240-1252. doi: 10.1111/head.13551. Epub 2019 May 9. PMID 31074005
- [Background] Nierenburg H, Rabany L, Lin T, Sharon R, Harris D, Ironi A, Wright P, Chuang L. Remote Electrical Neuromodulation (REN) for the Acute Treatment of Menstrual Migraine: a Retrospective Survey Study of Effectiveness and Tolerability. Pain Ther. 2021 Dec;10(2):1245-1253. doi: 10.1007/s40122-021-00276-7. Epub 2021 Jun 17. PMID 34138449
- [Background] Grosberg B, Rabany L, Lin T, Harris D, Vizel M, Ironi A, O'Carroll CP, Schim J. Safety and efficacy of remote electrical neuromodulation for the acute treatment of chronic migraine: an open-label study. Pain Rep. 2021 Oct 14;6(4):e966. doi: 10.1097/PR9.0000000000000966. eCollection 2021 Nov-Dec. PMID 34667919
- [Background] Hershey AD, Lin T, Gruper Y, Harris D, Ironi A, Berk T, Szperka CL, Berenson F. Remote electrical neuromodulation for acute treatment of migraine in adolescents. Headache. 2021 Feb;61(2):310-317. doi: 10.1111/head.14042. Epub 2020 Dec 21. PMID 33349920
- [Background] Tepper SJ, Lin T, Montal T, Ironi A, Dougherty C. Real-world Experience with Remote Electrical Neuromodulation in the Acute Treatment of Migraine. Pain Med. 2020 Dec 25;21(12):3522-3529. doi: 10.1093/pm/pnaa299. PMID 32935848
- [Background] Esparham A, Stark-Inbar A, Jekel L, Tamir S, Rabany L, Ironi A, Gautreaux J, Rao R. Acute Treatment of Migraine in Adolescents: Real-World Analysis of Remote Electrical Neuromodulation (REN). Pediatr Neurol. 2023 May;142:51-55. doi: 10.1016/j.pediatrneurol.2023.02.008. Epub 2023 Feb 21. PMID 36931109
- [Result] Ailani J, Rabany L, Tamir S, Ironi A, Starling A. Real-World Analysis of Remote Electrical Neuromodulation (REN) for the Acute Treatment of Migraine. Front Pain Res (Lausanne). 2022 Jan 18;2:753736. doi: 10.3389/fpain.2021.753736. eCollection 2021. PMID 35295483
- See also: Results for NCT05443659 — https://pubmed.ncbi.nlm.nih.gov/36931109/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nerivio Users Age 12-18: Adolecents with migraine who used theNerivio REN device for treating theitr migraine
Period: Overall Study
Arm/Group | Nerivio Users Age 12-18
Started | 1629
Completed | 1629
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adolescents with migraine who used the Nerivio REN device for treatment of their migraine
Groups:
- Nerivio Users Age 12-18: Adolecents with migraine who used the nerivio REN device for treating theitr migraine
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 1629
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participant at the day of creating a nerivio account Population: The age was calculated once per all study participants following by a subanalysis for each gender
  years
    Age, All | 15.9 (1.3)
    Age, female: number analyzed (Participants) | 1313
    Age, female | 15.8 (1.1)
    Age, Male: number analyzed (Participants) | 258
    Age, Male | 16.0 (1.7)
    Age, not identified: number analyzed (Participants) | 58
    Age, not identified | 16.1 (1.9)
Sex/Gender, Customized [Count of Participants; unit: Participants] — The gender of the participants (female, male, not identified)
  Participants
    Female | 1313
    Male | 258
    Not identifies | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Consistent Pain Relief at 2 Hours Post-treatment
Description: The proportion of subjects reporting pain relief at 2 hours post-treatment without the use of rescue medication in at least 50% of all their treatments. Pain relief is defined as an improvement from severe or moderate pain to mild or no pain, Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain)
Time Frame: 2 hours post treatment, up to 16 months from the 1st treatment
Population: REN users at the age of 12-=18 who used the Nerivio device as a single therapy (without rescue treatments were used) and had at least two evaluable treatments (with data at T=0h and T=2h) and repoerted baseline headache of moderate or severe in T=0h
Measure: Count of Participants; unit: Participants
Groups:
- Nerivio Users Age 12-18: Adolecents with migraine who used the nerivio REN device for treating their migraine and had reported the treatment questionnaire (both T=0h and T=2h) at least twice
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 262
Participants | 158

2. Secondary Outcome: Consistent Pain Freedom at 2 Hours Post-treatment
Description: The proportion of subjects reporting freedom from pain at 2 hours post-treatment without the use of rescue medication in at least 50% of all their treatments. Pain freedom is defined as reduction from severe or moderate or mild pain to no pain, Pain level is reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain,3- Severe pain)
Time Frame: 2 hours post treatment, up to 16 months from the 1st treatment
Population: REN users at the age of 12-18 who used the Nerivio device as a single therapy (without rescue treatments were used) and had at least two evaluable treatments (with data at T=0h and T=2h) and reported a type of headache in T=0h and no headache in the T=2h questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 289
Participants | 76

3. Secondary Outcome: Consistent Usage of Migraine Abortive (Rescue) Medications
Description: The proportion of subjects with REN treatments without the use of pharmacological migraine abortive (rescue) medication (either over the counter or prescribed), or with a combination of rescue medication or without any treatment at all at 2 hours post-treatment in at least 50% of all their treatments.
Time Frame: 2 hours post treatment, up to 16 months from the 1st treatment
Population: REN users at the age of 12-18 who used the Nerivio device as a single therapy (without rescue treatments were used) or with a combination of Nerivio and rescue medication or without any treatment at all and had at least two evaluable treatments (with data at T=0h and T=2h)
Measure: Count of Units; unit: Treatments with reportad medication
Units Other Than Participants: Treatments with reportad medication
Groups:
- Nerivio Treatments Performed by Users Aged 12-18: the number of nerivio treatments performed by adolecents with migraine who used the nerivio REN device for treating their migraine
Arm/Group | Nerivio Treatments Performed by Users Aged 12-18
Number analyzed (Participants) | 1629
Number analyzed (Treatments with reportad medication) | 2365
Treatments with reportad medication
  Treatments with Nerivio only | 1524
  Treatments with Nerivio and OTC medications | 439
  reatments with Nerivio andTriptan Rx | 180
  reatments with Nerivio and other Rx | 222

4. Secondary Outcome: Consistent Functional Disability Relief at 2 Hours Post-treatment
Description: The proportion of subjects reporting Functional Disability (FD) relief at 2 hours post-treatment without the use of rescue medication in at least 50% of all their treatments. FD relief is defined as an improvement from severe or moderate limitation to some or no limitation. FD level is reported using a 4-point Likert scale (0 - No limitation, 1 - Some limitation, 2 - Moderate limitation, 3 - Severe limitation)
Time Frame: 2 hours post treatment, up to 16 months from the 1st treatment
Population: REN users at the age of 12-18 who used the Nerivio device as a single therapy (without rescue treatments were used) and had at least two evaluable treatments (with data at T=0h and T=2h) and reported a reduction of at least one grade in the functional disability scale at T=2h
Measure: Count of Participants; unit: Participants
Groups:
- Nerivio Users Age 12-18: Adolecents with migraine who used the nerivio REN device for treating their migraine
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 255
Participants | 159

5. Secondary Outcome: Consistent Functional Disability Disappearance at 2 Hours Post-treatment
Description: The proportion of subjects reporting no Functional Disability (FD) at 2 hours post-treatment without the use of rescue medication in at least 50% of all their treatments. FD disappearance is defined as an improvement from severe or moderate or limitation to no limitation. FD level is reported using a 4-point Likert scale (0 - No limitation, 1 - Some limitation, 2 - Moderate limitation, 3 - Severe limitation).
Time Frame: 2 hours post treatment, up to 16 months from the 1st treatment
Population: REN users at the age of 12-18 who used the Nerivio device as a single therapy (without rescue treatments were used) and had at least two evaluable treatments (with data at T=0h and T=2h) and had a score of at least 1 in the functional disability scale and reported no functional disability at T=2h
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 255
Participants | 155

6. Other Pre Specified Outcome: Treatment Intensity Distribution
Description: The mean intensity of the stimulation collected for all treatments that were performed within the study
Time Frame: 45 minutes post treatment, up to 16 months from the 1st treatment
Population: Nerivio users at the age of 12-18 who treated at least once with the Nerivio device
Measure: Count of Units; unit: Nerivio treatments
Units Other Than Participants: Nerivio treatments
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 1629
Number analyzed (Nerivio treatments) | 13681
Nerivio treatments
  Intensity level 1-5 | 22
  Intensity level 6-10 | 250
  Intensity level 11-15 | 1678
  Intensity level 16-20 | 2274
  Intensity level 21-25 | 2492
  Intensity level 26-30 | 2203
  Intensity level 31-35 | 1661
  Intensity level 36-40 | 1033
  Intensity level 41-45 | 687
  Intensity level 46-50 | 529
  Intensity level 51-55 | 264
  Intensity level 56-60 | 210
  Intensity level 61-65 | 115
  Intensity level 66-70 | 79
  Intensity level 71-75 | 33
  Intensity level 76-80 | 38
  Intensity level 81-85 | 30
  Intensity level 86-90 | 29
  Intensity level 91-95 | 19
  tensity level 96-100 | 35

7. Other Pre Specified Outcome: Device Related Adverse Events
Description: Incidence of device-related adverse events reported by subjects
Time Frame: Up to 16 months
Population: Nerivio users at the age of 12-18 who used the device at least once
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Users Age 12-18
Number analyzed (Participants) | 1629
Participants | 3

ADVERSE EVENTS:
Time Frame: up to 18 months
Arm/Group | Nerivio Users Age 12-18
All-Cause Mortality (participants affected / at risk) | 0/1629
Serious Adverse Events (participants affected / at risk) | 0/1629
Other Adverse Events (participants affected / at risk) | 3/1629
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerivio Users Age 12-18 (N=1629)
Tingling (Skin and subcutaneous tissue disorders) | 2 (2)
Arm soreness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1. - this is not a controlled study. it has a single arm, of Nerivio users
2. - Efficacy and medication data were voluntarily provided by patients through the app, which contributed to the fact that not all adolescent users provided the required information at the beginning of the treatment and following two hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT05443659/Prot_SAP_000.pdf